CLINICAL TRIAL: NCT01056705
Title: The Phase Ⅱ Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains
Brief Title: The Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains (IPV)
Acronym: Sabin IPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); National Institute for the Control of Pharmaceutical and Biological Products, China (Other)
Responsible Party: Principal Investigator, Guoyang Liao, Head of Biologicals No.5, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: imbcams-02; SFDA2007L02021 (Other: China state food and drug adminstration)
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliomyelitis Vaccine; Sabin Strains; poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated; Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: Experiment Infants (Experimental): Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) formulation A. 3x0.5ml intramuscular injections;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Cohort 2: Experiment infants (Experimental): Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) formulation B. 3x0.5ml intramuscular injections;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Cohort 3: Experiment infants (Experimental): Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) formulation C. 3x0.5ml intramuscular injections;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Cohort 4: Experiment infants (Experimental): Biological: Oral Poliomyelitis Vaccine (OPV).3x0.1ml oral;
  Interventions: Biological: Oral Poliomyelitis Vaccine
- Cohort 5: Experiment infants (Experimental): Biological: Inactivated Poliomyelitis Vaccine (Salk strains). 3x0.5ml intramuscular injections;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Salk strains).

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — Inactivated Poliomyelitis Vaccine (Sabin strains) formulation A. 3x0.5ml intramuscular injections,one month apart.
  Other Names: Sabin IPV
  Arms: Cohort 1: Experiment Infants
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — Inactivated Poliomyelitis Vaccine (Sabin strains) formulation B. 3x0.5ml intramuscular injections, one month apart.
  Other Names: Sabin IPV
  Arms: Cohort 2: Experiment infants
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — Inactivated Poliomyelitis Vaccine (Sabin strains) formulation C. 3x0.5ml intramuscular injections, one month apart.
  Other Names: Sabin IPV
  Arms: Cohort 3: Experiment infants
Biological: Oral Poliomyelitis Vaccine — Oral Poliomyelitis Vaccine (OPV).3x0.5mloral, one month apart.
  Other Names: OPV
  Arms: Cohort 4: Experiment infants
Biological: Inactivated Poliomyelitis Vaccine (Salk strains). — 3x0.5ml intramuscular injections, one month apart.
  Other Names: Salk IPV
  Arms: Cohort 5: Experiment infants

SUMMARY:
Based on pre-clinical trial and phase 1 clinical data and principle of GCP, the objective of phase Ⅱ clinical trial is to evaluate safety and immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains(Sabin IPV).

DETAILED DESCRIPTION:
The Sabin IPV was manufactured with poliovirus type1, 2, 3 Sabin strains and Vero cells by microcarrier culture in 550 liter bioreactors. The virus suspension was harvested ,ultra-concentrated, purified and inactivated with formalin. Three formulations A,B,C of Sabin IPV were used, the DAg contents for A were type1 45,type2 64,type3 67.5 DU /0.5ml/per dose; for B 30,32,45 DU/0.5ml/per dose; for C 15,16,22.5 DU/0.5ml/per dose.

Oral Poliomyelitis Vaccine(OPV)was manufactured by Institute of Medical Biology, Chinese Academy of Medical Sciences.Trivalent OPV contains Polioviruses Type 1 6.0 log CCID Type 2 5.0 log Type 3 5.5log /0.1ml/per dose Inactivated Poliomyelitis Vaccine (Salk strains)was manufactured by Sanofi Pasteur DAg contents /0.5ml/per dose were Type 1 40 DU,Type 2 8DU,Type 3 32DU.

This is a randomized, blind phase 2 clinical trial. Total 500 infants (ages 60 days to 90 days) were selected , randomized to five groups(each group n=100) Sabin IPV formulations A,B,C,OPV ,Salk IPV were separately given to each group with three doses one month apart respectively.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age from 60 days to 90 days;
* Adults, parent(s) or guardians are able to understand and sign informed consent for participation;
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions;
* Infants no vaccinated with poliovaccine or other preventive biologicals in recent 7 days;
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Have medical record of participants or their family on allergy, convulsion, falling sickness, encephalopathy and psychopathy;
* Low platelet or bleeding disorder do not allow vaccination into the muscle;
* Have damaged or lower immunological function;
* Received blood, plasma or immunoglobulin treatment since birth;
* Have inborn abnormality, develop obstacles or clinical diagnostic serious chronic ( Down Syndrome, diabetes, sickle cell anemia or neural Guillain-Barre Syndrome );
* Have or be doubtful of following diseases: respiratory system diseases, acute infection or active chronic, cardiovascular diseases, liver and kidney diseases, skin diseases, HIV.

Exclusion Criteria for doses 2 and 3

* Have serious anaphylaxis or high fever, convulsion during first dose;
* Have any circus of Exclusion Criteria after Eligible for study;
* Have serious adverse event which related to previous vaccination; Withdrawal and Discontinuance Criteria;
* Received necessary or interference study drugs such as: immune-inhibition or immune-stimulating agents;
* Vaccinated with any other vaccine（except DTP）;
* Stop observation determined by investigator owing to occurring serious adverse event;

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains by different does on Healthy infants . | one year

CONTACTS AND LOCATIONS:
Overall Officials: Liao Guoyang, PHD, Principal Investigator — Institute of Medical Biology, Chinese Academy of Medical Sciences; Li Rongcheng, MD, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control; Li Changgui, PHD, Principal Investigator — National Institute for the Control of Pharmaceutical and Biological Products, China
Locations (1):
- Pingle Center for Disease Control and Prevention, Pingle County, Guangxi, China

REFERENCES:
- [Derived] Sun M, Li C, Xu W, Liao G, Li R, Zhou J, Li Y, Cai W, Yan D, Che Y, Ying Z, Wang J, Yang H, Ma Y, Ma L, Ji G, Shi L, Jiang S, Li Q. Immune Serum From Sabin Inactivated Poliovirus Vaccine Immunization Neutralizes Multiple Individual Wild and Vaccine-Derived Polioviruses. Clin Infect Dis. 2017 May 15;64(10):1317-1325. doi: 10.1093/cid/cix110. PMID 28419204
- [Derived] Liao G, Li R, Li C, Sun M, Li Y, Chu J, Jiang S, Li Q. Safety and immunogenicity of inactivated poliovirus vaccine made from Sabin strains: a phase II, randomized, positive-controlled trial. J Infect Dis. 2012 Jan 15;205(2):237-43. doi: 10.1093/infdis/jir723. Epub 2011 Dec 8. PMID 22158682